CLINICAL TRIAL: NCT06770166
Title: The Effect of Chamomile on Healing After Tooth Extraction: a Retrospective Randomized Controlled Trial
Brief Title: The Effect of Chamomile on Healing After Tooth Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: reyhansaglam (Other)
Responsible Party: Sponsor-Investigator, reyhansaglam, PhD, Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 10840098-604.01.01-21824
Record Dates: First submitted 2025-01-06; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Tooth Extraction Status Nos
Keywords: chamomile; chlorhexidine; tooth extraction

STUDY DESIGN:
Intervention Model Description: A prospective randomized controlled clinical trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- physiological serum mouthwash group (control group) (Active Comparator): After extraction, 40 patients were given saline mouthwash to use for 7 days.
  Interventions: Other: Physiological serum mouthwash
- chlorhexidine mouthwash group (Active Comparator): After extraction, 40 patients were given chlorhexidine mouthwash to use for 7 days.
  Interventions: Other: Chlorhexidine mouthwash
- chamomile mouthwash group (Active Comparator): After extraction, 40 patients were given chamomile mouthwash to use for 7 days.
  Interventions: Other: Chamomile mouthwash

INTERVENTIONS:
Other: Physiological serum mouthwash — Physiological serum contains sodium chloride : 0.009 g/ml, sodium 154 (mEq/I), chloride 154 (mEq/I)].
  Arms: physiological serum mouthwash group (control group)
Other: Chlorhexidine mouthwash — Chlorhexidine mouthwash contains 0.12% chlorhexidine digluconate and 0.15% benzydamine hydrochloride.
  Arms: chlorhexidine mouthwash group
Other: Chamomile mouthwash — Chamomile mouthwash contains 10% chamomile in physiological serum.
  Arms: chamomile mouthwash group

SUMMARY:
After impacted wisdom tooth extraction, patients frequently complain of pain, edema, and limited mouth opening. After the procedure, patients are routinely recommended to use chlorhexidine and physiological serum-based mouthwashes. The antibacterial and anti-inflammatory effects of warm chamomile tea have been reported in the literature. In addition, the neuroprotective, antiallergic, antioxidant, antiseptic and spasmolytic properties of chamomile have been reported. The aim was to compare the effects of these gargles in terms of pain, mouth opening, burning sensation in the mouth, edema, and discoloration of the tongue and teeth.

DETAILED DESCRIPTION:
The study was planned to be applied to 120 patients, 40 in each group. In the ASA 1 group, the mouth opening of the patients was recorded before the tooth extraction procedure. Impacted teeth were extracted using Ultracain D-S Forte (Articaine HCl: 40mg/ml, Epinephrine HCl: 0.012 mg/ml) as a local anesthetic. Dental units were prepared under sterile conditions. The patients were covered with a sterile drape. The lower wisdom tooth was extracted with open (surgical) extraction. The mucoperisoteal flap was lifted with a number 15 surgical scalpel, and the tooth was extracted using round and fissure-tipped steel burs with a handpiece. After tooth extraction, if there was granulation tissue in the extraction socket, it was curetted and irrigated with physiological serum [sodium chloride: 0.009 g/ml, sodium 154 (mEq/I), chloride 154 (mEq/I)]. After bleeding control, patients were given written and verbal postoperative advice. Antibiotics and analgesics were prescribed to patients, chlorhexidine gargle was recommended to 30 patients, saline gargle to 30 patients, and chamomile tea gargle to 30 patients. Patients were given VAS pain scores, numbered 0-10, to record for 7 days after extraction. Patients were called back to the clinic on the 2nd and 7th days after tooth extraction to assess pain, burning sensation and color change in the tongue, mouth opening, and edema. Sutures were removed on the 7th postoperative day.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status I patients,
2. did not have the medical history of being allergic to local anesthesia
3. did not have the medical history of being allergic to CHX,
4. did not have acute infection at the tooth area
5. absence of any pathology at the area.

Exclusion Criteria:

1. Participants with medically compromised condition,
2. pregnant females
3. smokers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2024-10-26 (Actual); Study Completion 2024-10-26 (Actual)

PRIMARY OUTCOMES:
Patients pain value | The patient marked the pain value every day for one week.
  visual analog scale (VAS) is used for pain assessment. The patient marked the pain value on the 0-10 visual analog scale.
maximum mouth opening | maximum mouth opening was measured preoperatively, postoperative 3rd and 7th days.
  maximum mouth openin were measured with the reference of 11 and 41 teeth. are used for interincisal distances

CONTACTS AND LOCATIONS:
Overall Officials: reyhan saglam, PhD, Principal Investigator — İstanbul Medipol university
Locations (1):
- Istanbul Medipol University Dental School, Istanbul, Unkapani, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No